CLINICAL TRIAL: NCT04710277
Title: Randomized Controlled Trial of a Novel Multimodal Pain Control Protocol for Minimally Invasive Gynecologic Surgery
Brief Title: Novel Multimodal Pain Control Protocol for Minimally Invasive Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Silpa Nekkanti, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020H0077
Record Dates: First submitted 2020-12-29; First posted 2021-01-14 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Pain; Narcotic Use; Cryotherapy Effect
MeSH Terms: conditions — Pain, Postoperative | interventions — Ice; Cryotherapy

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned prospectively to one of two interventions according to protocol to evaluate the effect of the intervention on their postoperative pain, quality of recovery, patient satisfaction, and overall analgesic use.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel multimodal protocol group (Experimental): They will receive scheduled topical ice therapy for 24 hours after surgery. It will be applied over abdominal incisions for 20 minutes every 2-3 hours. Acetaminophen and an NSAID will be scheduled for 96 hours. While inpatient, they will receive acetaminophen 975 mg every 8 hours and IV Toradol 15-30 mg every 6 hours with change to ibuprofen 800 mg every 8 hours when tolerating oral intake. They may take oxycodone 5 mg every 4-6 hours as needed (PRN) for breakthrough pain and pain score >6. They may use ice PRN after 24 hours. They will be prescribed acetaminophen 1000 mg every 8 hours and ibuprofen 800 mg every 8 hours for 96 hours postoperative. They may take them as needed after. If the participant used 0 narcotics in the first 24 hours, they will not be prescribed a narcotic. If up to 5 tablets were used, they will be prescribed 5 tablets of oxycodone 5 mg every 6 hours PRN. If more than 5 tablets were used, they will be prescribed 10 tablets of oxycodone 5 mg every 6 hours PRN.
  Interventions: Other: Opioid-sparing multimodal pain management
- Usual care protocol group (Active Comparator): Participants randomly assigned to the usual care protocol will receive current standard of care: scheduled acetaminophen and an NSAID for 24 hours. They will take acetaminophen 975 mg every 8 hours. They will also receive IV toradol 15 to 30 mg every 6 hours then switch to ibuprofen 800 mg every 8 hours when tolerating oral intake. They can also take oxycodone 5 mg every 4 to 6 hours on an as needed (PRN) basis for breakthrough pain with a pain score >6. Per our current standard of care, usual care participants will be allowed to use either topical heat or ice on an as needed basis during their recovery. On discharge home, they will be prescribed acetaminophen 1000 mg every 8 hours PRN and ibuprofen 800 mg every 8 hours PRN. They will also be prescribed 15 tablets of oxycodone 5 mg every 6 hours PRN.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Opioid-sparing multimodal pain management — Ice pack applied to abdominal incisions for 20 minutes every 2 to 3 hours for 24 hours after surgery and scheduled acetaminophen and NSAID for 96 hours after surgery. Narcotic pain medication for severe breakthrough pain.
  Other Names: Ice therapy; Ice pack; Cryotherapy
  Arms: Novel multimodal protocol group
Other: Usual care — Scheduled acetaminophen and NSAID for 24 hours after surgery. Narcotic pain medication for severe breakthrough pain.
  Arms: Usual care protocol group

SUMMARY:
The study is a randomized controlled trial investigating a multimodal postoperative pain management protocol which will include use of ice therapy and scheduled opioid-sparing medications for pain control after minimally invasive gynecologic surgery.

DETAILED DESCRIPTION:
The study is a randomized controlled trial investigating a multimodal postoperative pain management protocol which will include use of ice therapy and scheduled opioid-sparing medications for pain control after minimally invasive gynecologic surgery. The study will include women >/= 18yo who speak English and are admitted for observation after a qualifying laparoscopic or robotic gynecologic procedure. The investigators will identify potential participants from the operating schedule, screen for any exclusion criteria, and approach those eligible for inclusion on the day of surgery. All participants will receive a pain regimen with medications commonly used to manage post-surgical pain including nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen, and prescription opioids. Participants randomized to the intervention arm will receive prolonged scheduled NSAID and acetaminophen (96 hours instead of 24 hours) and will receive 24 hours of intermittent ice-therapy (20 minutes every 2-3 hours) on their abdominal incisions beginning within 1-2 hours after surgery. On post-operative day or day 1, a study investigator will administer a study questionnaire to all participants which will include a pain score, satisfaction score, and quality of recovery validated survey (the QoR-40). After discharge, participants will complete short web-based survey questionnaires on day 2 and 3. On day 4 a final and more comprehensive web-based survey will be sent to all participants which will include the 24-hour assessment in addition to the QoR-40 questionnaire, a final satisfaction questionnaire, and pill counts of left-over discharge medications. The day 4 survey completes the participants active part in the study. On or after day 30 a chart review will be performed to assess for post-operative complications, emergency room visits, telephone calls, unexpected office visits, and refill requests. An Ohio Rx Reporting System (OARRS) report will further screen for any additional narcotic prescriptions in the 30 day postoperative period. This will mark completion of participation in study. The completion of the study questionnaires is anticipated to take about 1.5 to 2 hours in total time throughout the study. There are no additional clinic visits or costs associated with participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Minimally invasive (laparoscopic or robotic) major gynecologic procedures including: pelvic floor procedures (uterosacral ligament suspension, sacrocolpopexy, Burch colposuspension) with or without concomitant hysterectomy, adnexal surgery, or vaginal surgery; total or supracervical hysterectomy with or without concomitant adnexal surgery, vaginal surgery, or other minor gynecologic procedures
* Patients admitted to the hospital for at least an overnight observation after their surgery
* English-speaking
* Surgery being performed by one of the five attending surgeons included in study

Exclusion Criteria:

* Pregnancy. If patient is of childbearing potential and not using contraception a urine pregnancy test will be completed as part of standard practice as part of pre-operative labs.
* Diagnosis of chronic pelvic pain. Documented pelvic pain noted to be of >6 months duration.
* Diagnosis or history of chronic opioid use. Defined as use of opioids most days, for more than 3 months.
* Diagnosis or history of opioid abuse disorder.
* Current daily opioid use.
* Liver, renal, or cardiac disease that is/are a contraindication to any medications used in the study.
* Allergy or intolerance to any medication used in the study (with exception of oxycodone which can be substituted for hydromorphone if necessary).
* Dementia or inability to understand or respond to the study measurement tools.
* Intraoperative exclusion criteria (to be reviewed after surgery is complete): conversion to total vaginal procedure or laparotomy, major intraoperative complications that would deem participant inappropriate for trial (hemorrhage, blood transfusion, conversion to laparotomy, bowel surgery, major urologic procedures including bladder or ureteral repair).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Day 1 pain score assessed by NRS-11 | During the intervention on postoperative day 1 between 0600 to 0900
  Postoperative day 1 or Day 1 pain score will be measured using a commonly used and validated 11-point numerical rating scale (NRS-11) for pain intensity the morning after surgery between 0600 to 0900. The patient will be prompted to evaluate their current pain at rest. A score of zero will correspond with "no pain" and a score of 10 corresponds with "worst possible pain." The outcome will be recorded directly into their Day 1 study survey in REDCap.

SECONDARY OUTCOMES:
Day 2 to 4 pain score assessed by NRS-11 | During the intervention on postoperative day 2 to 4
  Pain scores on Day 2, 3, and 4: An NRS-11 pain score at rest will be collected on Day 2, 3, and 4 via electronic REDCap survey. A score of zero will correspond with "no pain" and a score of 10 corresponds with "worst possible pain."
Quality of Recovery assessed by QoR-40 | During the intervention on postoperative day 1 and 4
  Participants will be asked to complete a validated quality of recovery questionnaire (the QoR-40) on Day 1 in AM as part of their Day 1 study survey that will be administered electronically directly into REDCap. The QoR-40 will also be administered on Day 4 via electronic REDCap survey. QoR-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).
Patient satisfaction with pain control assessed by NRS-11 | During the intervention on postoperative day 1 and 4
  Participants will be asked to rate their post-operative pain control satisfaction using an NRS-11 scale for satisfaction. The question prompt on Day 1 will read "On a scale of 0 to 10 how would you rate your satisfaction with your postoperative pain control in the last 24 hours?" A score of 0 corresponds with "very dissatisfied" and a score of 10 corresponds with "very satisfied." A pain control satisfaction NRS-11 will also be administered on Day 4 as part of the electronic REDCap survey. The question prompt on Day 4 will read "On a scale of 0 to 10 how would you rate your satisfaction with your postoperative pain control since you left the hospital?"
Patient satisfaction with ice therapy assessed by NRS-11 | During the intervention on postoperative day 1 and 4
  Patient satisfaction with the scheduled 24 hour ice therapy will be assessed using the same NRS-11 satisfaction scale as described above. Ice therapy satisfaction will be assessed on Day 1 as part of the Day 1 AM REDCap survey to be administered electronically directly into REDCap. The question prompt with the NRS-11 will read "On a scale from 0 to 10, how would you rate your satisfaction with the ice therapy as part of your postoperative pain regimen?" A score of 0 corresponds with "very dissatisfied" and a score of 10 corresponds with "very satisfied." We will also ask the following non-validated questions aimed at assessing patient satisfaction with their ice therapy: "Did you feel that the ice therapy was helpful? Did you feel that the ice therapy was bothersome? If you had to do it over, would you use the ice therapy again?" These same questions will be administered as part of the Day 4 electronic REDCap survey.
Patient satisfaction with ice therapy assessed by brief questionnaire | During the intervention on postoperative day 1 and 4
  Patient satisfaction with the scheduled 24 hour ice therapy will also be assessed by asking a brief questionnaire including the following non-validated questions: "Did you feel that the ice therapy was helpful? Did you feel that the ice therapy was bothersome? If you had to do it over, would you use the ice therapy again?" The answer options will be "yes" or "no". These same questions will be administered as part of the Day 4 electronic REDCap survey.
Analgesic use - opioids measured by morphine equivalents | Immediately after the surgery from postoperative day 0 to 4
  Administration or use of any opioids will be extracted from the medical record and recorded in the study database for the pre-operative, intraoperative, immediate post-operative (i.e. PACU), and inpatient time points. Any use of intravenous opioids will be specifically noted in study database. Once discharged from the hospital, participants will be asked to fill out a daily pain control and medication use electronic survey on Day 2, 3, and 4. The brief survey will have fields for frequency and dosage in milligrams of opioid use over the past 24 hours. All opioid information will be converted into oral morphine equivalents using an equianalgesic dosage conversion calculator.
Analgesic use frequency - acetaminophen | Immediately after the surgery from postoperative day 0 to 4
  Administration or use of acetaminophen will be extracted from the medical record and recorded in the study database for the pre-operative, intraoperative, immediate post-operative (i.e. PACU), and inpatient time points. Once discharged from the hospital, participants will be asked to fill out a daily pain control and medication use electronic survey on Day 2, 3, and 4. The brief survey will have a field for frequency of acetaminophen use with the ability to select from the following options: "every 4 hours, every 6 hours, every 8 hours, twice a day, once a day, or other".
Analgesic use dosage - acetaminophen measured by milligrams | Immediately after the surgery from postoperative day 0 to 4
  Administration or use of acetaminophen will be extracted from the medical record and recorded in the study database for the pre-operative, intraoperative, immediate post-operative (i.e. PACU), and inpatient time points. Once discharged from the hospital, participants will be asked to fill out a daily pain control and medication use electronic survey on Day 2, 3, and 4. The brief survey will ask dosage of acetaminophen use measured in milligrams over the past 24 hours.
Analgesic use frequency - NSAID | Immediately after the surgery from postoperative day 0 to 4
  Administration or use of any NSAID will be extracted from the medical record and recorded in the study database for the pre-operative, intraoperative, immediate post-operative (i.e. PACU), and inpatient time points. Once discharged from the hospital, participants will be asked to fill out a daily pain control and medication use electronic survey on Day 2, 3, and 4. The brief survey will have a field for frequency of NSAID use with the ability to select from the following options: "every 4 hours, every 6 hours, every 8 hours, twice a day, once a day, or other".
Analgesic use dosage - NSAID measured by milligrams | Immediately after the surgery from postoperative day 0 to 4
  Administration or use of any NSAID will be extracted from the medical record and recorded in the study database for the pre-operative, intraoperative, immediate post-operative (i.e. PACU), and inpatient time points. Once discharged from the hospital, participants will be asked to fill out a daily pain control and medication use electronic survey on Day 2, 3, and 4. The brief survey will ask dosage of NSAID use measured in milligrams over the past 24 hours.
Analgesic use - other neuraxial agent | Immediately after the surgery from postoperative day 0 to 4
  Administration or use of any other neuraxial agent or medication for pain (i.e. gabapentin) will be extracted from the medical record and recorded in the study database for the pre-operative, intraoperative, immediate post-operative (i.e. PACU), and inpatient time points. Once discharged from the hospital, participants will be asked to fill out a daily pain control and medication use electronic survey on Day 2, 3, and 4. The brief survey will have a "free text" field to allow the participant to describe any use of a medication for pain not listed above.
Ice therapy use frequency | Immediately after the surgery from postoperative day 0 to 4
  Administration or use of ice therapy will be extracted from the nurse ice administration logs. This will be recorded in the study database for the pre-operative, intraoperative, immediate post-operative (i.e. PACU), and inpatient time points. Once discharged from the hospital, participants will be asked to fill out a daily pain control and medication use electronic survey on Day 2, 3, and 4. The brief survey will have fields for frequency of ice therapy with the ability to select from the following options: "every 1-2 hours, every 2-3 hours, every 3-4 hours, every 4-5 hours, every 5-6 hours, every 6-8 hours, every 8-12 hours, or once".
30-day postoperative outcomes | After the surgery on postoperative day 1 to 30
  After Day 30, a study investigator will perform a chart review and an OARRS (Ohio automated Rx reporting system) report on each participant in order to complete the secondary outcomes of 30-day post-operative complications, unexpected office phone calls or visits, emergency room visits, readmissions, and medication refill requests.
Adverse events (AEs) | During the intervention on postoperative day 1 to 4
  Throughout the study we will monitor for AEs, both anticipated and unanticipated. Possible AEs for scheduled ice therapy could include local discomfort, skin irritation, or ice burn if used incorrectly without a barrier between ice therapy and skin. Ice therapy side effects or AEs will be directly queried on Day 1 by study investigator, and on Day 2, 3, and 4 via electronic survey. All AEs will be reported to The Ohio State IRB according to the reporting guidelines. AEs will be assessed at each clinical/research visit and reported with study outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Silpa Nekkanti, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No